CLINICAL TRIAL: NCT02118545
Title: Preoperative Von Willebrand Factor to Predict Postoperative Liver Dysfunction and Morbidity After Liver Resection
Brief Title: Von Willebrand Factor to Predict Postoperative Outcome
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Patrick Starlinger, MD, PhD, Medical University of Vienna
Other Study IDs: Vie-Sal-Ber
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2015-09

CONDITIONS: Liver Dysfunction; Morbidity; Mortality; Hospitalisation
Keywords: vWF; Liver Resection; Liver Dysfunction; Liver Regeneration; Postoperative Outcome
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- vWF and postoperative Outcome: An independent prospective validation cohorts will be obtained from 4 different Institutions: 2 in Vienna , 1 in Salzburg and 1 in Bern

SUMMARY:
vWF is stored in weibel-palade-bodies of endothelial cells as well as alpha-granula of platelets and is released upon their activation. Endothelial cell dysfunction as well as platelet activation often occur in liver disease and portal hypertension, which may lead to an increase in circulating vWF levels. Indeed, multiple studies have reported that liver disease is associated with increased circulating vWF- antigen (vWF-Ag). Furthermore, increased circulating vWF -Ag Levels have been shown to be associated with increased mortality rates in patients with chronic liver disease. Within a prospective evaluation cohort, the investigators were able to document that patients with increased vWF-Ag levels prior to liver resection suffered from an increased incidence of postoperative liver dysfunction and morbidity. Within this prospective multicenter validation study, the investigators now aim to prospectively validate that circulating vWF-Ag prior to liver resection is a valuable marker to predict postoperative clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing liver resection
* only patients with either hepatocellular carcinoma, cholangiocellular carcinoma or colorectal cancer liver metastasis will be included

Exclusion Criteria:

* inherited coagulopathy
* age > 85

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver resections for either hepatocellular carcinoma, cholangiocellular carcinoma or colorectal cancer liver metastasis. vWF-Ag will be evaluated prior to liver resection
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Postoperative Liver Dysfunction | 90 postoperative days
  Preoperative vWF-Ag Predicts Postoperative Liver Dysfunction after Liver Resection

SECONDARY OUTCOMES:
Number of Participants with Postoperative Morbidity | 90 postoperative days
  Preoperative vWF-Ag Predicts Postoperative Morbidity after Liver Resection
Number of Participants with Postoperative Mortality | 90 postoperative days
  Preoperative vWF-Ag Predicts Postoperative Mortality after Liver Resection
Days of Postoperative Hospitalisation | 90 postoperative days
  Preoperative vWF-Ag Predicts Postoperative Hospitalisation after Liver Resection

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Starlinger, MD, PhD, Principal Investigator — Medical University Vienna; Thomas Gruenberger, MD, Study Chair — Rudolf Foundation Clinic; Stefan Stättner, MD, Study Chair — Paracelsus Medical University; Guido Beldi, MD, Study Chair — University of Bern
Locations (4):
- Austria (3):
  - Medical University Vienna, Vienna, Vienna
  - Paracelsus Medical University, Salzburg
  - Rudolf Foundation Clinic, Vienna
- University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Starlinger P, Pereyra D, Haegele S, Braeuer P, Oehlberger L, Primavesi F, Kohler A, Offensperger F, Reiberger T, Ferlitsch A, Messner B, Beldi G, Staettner S, Brostjan C, Gruenberger T. Perioperative von Willebrand factor dynamics are associated with liver regeneration and predict outcome after liver resection. Hepatology. 2018 Apr;67(4):1516-1530. doi: 10.1002/hep.29651. Epub 2018 Feb 27. PMID 29140542